CLINICAL TRIAL: NCT06636162
Title: Early Phase 1 Window of Opportunity Study of Oral DSP-0390 in Grade II and III Gliomas
Brief Title: Window of Opportunity Study of DSP-0390 in Gliomas
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Sumitomo Pharmaceuticals America (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202412002
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Glioma, Malignant; Grade II Glioma; IDH Mutation
Keywords: Grade III Glioma; DSP-0390; IDH-mutant glioma; brain tumor; brain cancer
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Ten patients will be enrolled and treated with DSP-0390, and if the patients tolerate dosing well, another ten patients will be enrolled and treated with a higher dose of DSP-0390.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DSP-0390 120 mg (Experimental): The first 10 patients will be assigned to DSP-0390 120 mg once daily by mouth for approximately 2 weeks and up to 17 days prior to surgical resection, with the final dose being administered the morning of surgery.
  Interventions: Drug: DSP-0390
- DSP-0390 240 mg (Experimental): The next 10 patients will be assigned to DSP-0390 240 mg once daily by mouth for approximately 2 weeks and up to 17 days prior to surgical resection, with the final dose being administered the morning of surgery.
  Interventions: Drug: DSP-0390

INTERVENTIONS:
Drug: DSP-0390 — DSP-0390 will be administered orally with preferably 200 mL of water, or approximately one-half cup water. The patient will take DSP-0390 after a minimum of a 6-hour fast and will fast for 1 hour after taking the dose.

SUMMARY:
This study focuses on determining the pharmacokinetic and pharmacodynamic effect of DSP-0390 in brain and blood from patients with IDH-mutant WHO grade II or III glioma undergoing tumor resection. Tissue will be collected during surgical resection. Blood will be drawn at various time points throughout the 2 weeks of treatment. The hypothesis is that DSP-0390 will accumulate in brain tumor tissue at pharmacologically relevant concentrations, and that alterations in cholesterol metabolism driven by mutant IDH will increase susceptibility to DSP-0390 and lead to tumor cell death.

ELIGIBILITY:
Inclusion Criteria

* Either newly diagnosied, suspected lower grade glioma per radiographic features, or radiographic recurrence of a histologically confirmed grade II or III IDH-mutant glioma.
* Patient must be a candidate for surgical resection
* At least 18 years of age.
* Karnofsky ≥ 70%
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm (patient may not use G-CSF or GM-CSF to achieve this ANC level)
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9 g/dL (patient may not receive transfusion or use erythropoietin to obtain this Hgb level)
  * Total bilirubin ≤ 1.5 x IULN (or ≤ 3 x IULN for patients with known Gilbert's syndrome)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * International normalized ratio (INR), prothrombin time (PT), partial thromboplastin time (PTT), or activated partial thromboplastin time (aPTT) ≤1.5 x ULN. The use of anticoagulants is permitted as long as the PT/(a)PTT is within therapeutic limits (according to the local institution standard) and the patient has been on a stable anticoagulant regimen for at least 2 weeks prior to Day 1.
  * Creatinine Clearance of ≥40 mL/min per Cockroft-Gault formula or by a 24 hour urine.
* If a patient is using an antiepileptic medication, the patient is on a stable dose and without seizures for 14 days prior to Day 1. The antiepileptic medication used must not fall under any prohibited therapy category as defined in the protocol.
* If the patient is receiving corticosteroids at baseline, the dose administered is stable or decreasing for at least 5 days prior to Day 1. A higher stable dose of corticosteroids, if used as hormone replacement therapy, may be allowed upon discussion with the sponsor-investigator.
* The effects of DSP-0390 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (2 forms of acceptable contraception, including one barrier method) prior to study entry, for the duration of study participation, and for 6 months after the last dose of DSP-0390. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria

* Patient has had prior therapy with bevacizumab or other anti-vascular endothelial growth factor (VEGF) treatments within 3 months prior to Day 1.
* Patient has multifocal disease, leptomeningeal metastasis, or extracranial metastasis.
* Patient has a clinically significant abnormal ECG, including those where QT prolongation is determined by the Fridericia formula (QTcF >450 msec for males and >470 msec for females); and/or the patient has a history of Torsade de Pointes.
* Patient is known to have dysphagia, short-gut syndrome, gastroparesis, or other condition that may limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Patient is known to have active Crohn's or other inflammatory bowel disease.
* A history of other malignancy for which all treatment was completed at least 2 years before Day 1 and the patient has no evidence of disease. Exceptions include non-melanoma skin cancer, cervical carcinoma in situ, and superficial bladder cancer that has been removed or curatively treated.
* On active treatment for other, unrelated malignancy or currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to DSP-0390.
* Patient has taken concurrent use of prohibited medications: carbamazepine, phenytoin, phenobarbital, and other strong or moderate CYP3A4 inhibitors or inducers, and strong CYP2D6 inhibitors within 1 week or 5 half-lives (whichever is greater) prior to Day 1 or expects to use them during the study. Note both oral and IV ondansetron at doses ≤ 8mg q6 hours are permitted.
* The presence of any active retinal abnormality determined by screening ophthalmologic examination.
* Patient has significant cardiovascular disease, including New York Heart Association (NYHA) Class III or IV congestive heart failure, myocardial infarction, unstable angina, pectoris, clinically significant cardiac arrhythmias, or stroke in the preceding 6 months prior to Day 1.
* Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements, disorders associated with significant immunocompromised state, or ongoing or active infection.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of DSP-0390.
* Patients with HIV are eligible unless their CD4+ T-cell counts are <350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended, as long as the ART agents do not fall under exclusion #8.
* Patient has a known detectable viral load for hepatitis C, or evidence of a hepatitis B surface antigen.
* Patient has had a major non-neurologic surgical procedure, surgical resection, open biopsy, or significant traumatic injury within 4 weeks prior to Day 1 or anticipates needing a major surgical procedure during the course of the study.
* Patient has had a minor surgical procedure, fine needle aspirations, or core biopsies within 7 days prior to Day 1.
* Patient has received chemotherapy or investigational anticancer therapy within 4 weeks (except 6 weeks for nitrosoureas and immunotherapy, or 8 weeks for an implanted nitrosoureas wafer) prior to Day 1.
* Patient has had radiotherapy within 12 weeks prior to Day 1, unless relapse is confirmed by tumor biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Unbound DSP-0390 concentration in non-enhancing tumor tissue | At time of surgery following treatment (estimated to be 2 weeks)
  Unbound DSP-0390 concentration in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Changes in DSP-0390 concentration in plasma | From start of treatment through end of treatment (estimated to be 2 weeks)
  Unbound DSP-0390 concentration in plasma will be quantified using blood samples taken throughout treatment.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | From start of treatment through 30 day follow-up (estimated to be 6 weeks)
  Assessed using CTCAE v5.0
Incidence of grade 3 or higher study drug related adverse events (AEs) | From start of treatment through 30 day follow-up (estimated to be 6 weeks)
  Assessed using CTCAE v5.0
Lathosterol levels in non-enhancing tumor tissue | At time of surgery following treatment (estimated to be 2 weeks)
  Lathosterol levels in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Changes in lathosterol levels in non-enhancing tumor tissue | Baseline and at time of surgery following treatment (estimated to be 2 weeks)
  Lathosterol levels in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Zymostenol levels in non-enhancing tumor tissue | At time of surgery following treatment (estimated to be 2 weeks)
  Zymostenol levels in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Changes in zymostenol levels in non-enhancing tumor tissue | Baseline and at time of surgery following treatment (estimated to be 2 weeks)
  Zymostenol levels in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Lathosterol/zymostenol (L/Z) ratio in non-enhancing tumor tissue | At time of surgery following treatment (estimated to be 2 weeks)
  L/Z ratio in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Changes in lathosterol/zymostenol (L/Z) ratio in non-enhancing tumor tissue | Baseline and at time of surgery following treatment (estimated to be 2 weeks)
  L/Z ratio in non-enhancing tumor tissue will be quantified using tissue removed during resection after treatment.
Changes in lathosterol levels in blood | From start of treatment through 5 days of treatment
  Change in lathosterol levels in blood will be quantified after 5 days of DSP-0390 dosing.
Changes in lathosterol levels in blood | From start of treatment through 10 days of treatment
  Change in lathosterol levels in blood will be quantified after 10 days of DSP-0390 dosing.
Changes in lathosterol levels in blood | From start of treatment through 11 days of treatment
  Change in lathosterol levels in blood will be quantified after 11 days of DSP-0390 dosing.
Changes in lathosterol levels in blood | From start of treatment through day 15
  Change in lathosterol levels in blood will be quantified after 15 days of DSP-0390 dosing.
Changes in lathosterol levels in blood | From start of treatment through day 16
  Change in lathosterol levels in blood will be quantified after surgical resection.
Changes in zymostenol levels in blood | From start of treatment through 5 days of treatment
  Change in zymostenol levels in blood will be quantified after 5 days of DSP-0390 dosing.
Changes in zymostenol levels in blood | From start of treatment through 10 days of treatment
  Change in zymostenol levels in blood will be quantified after 10 days of DSP-0390 dosing.
Changes in zymostenol levels in blood | From start of treatment through 11 days of treatment
  Change in zymostenol levels in blood will be quantified after 11 days of DSP-0390 dosing.
Changes in zymostenol levels in blood | From start of treatment through day 15
  Change in zymostenol levels in blood will be quantified after 15 days of DSP-0390 dosing.
Changes in zymostenol levels in blood | From start of treatment through day 16
  Change in zymostenol levels in blood will be quantified after surgical resection.
Changes in L/Z ratio in blood | From start of treatment through 5 days of treatment
  Change in L/Z ratio in blood will be quantified after 5 days of DSP-0390 dosing.
Changes in L/Z ratio in blood | From start of treatment through 10 days of treatment
  Change in L/Z ratio in blood will be quantified after 10 days of DSP-0390 dosing.
Changes in L/Z ratio in blood | From start of treatment through 11 days of treatment
  Change in L/Z ratio in blood will be quantified after 11 days of DSP-0390 dosing.
Changes in L/Z ratio in blood | From start of treatment through day 15
  Change in L/Z ratio in blood will be quantified after 15 days of DSP-0390 dosing.
Changes in L/Z ratio in blood | From start of treatment through day 16
  Change in L/Z ratio in blood will be quantified after surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Omar H Butt, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu